CLINICAL TRIAL: NCT06515496
Title: A Clinical Trial to Examine the Efficacy of a Dietary Supplement to Improve the Health and Appearance of Hair.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scale Media Inc (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20413
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Hair Thinning; Hair Shedding
Keywords: Hair growth; Female pattern hair loss; Hair health
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in this arm will take the Scale HLV Clinical Formula Hair Vitamins.
  Interventions: Dietary Supplement: Scale HLV Clinical Formula Hair Vitamins
- Placebo (Placebo Comparator): Participants in this arm will take a placebo product consisting of rice flour in vegetable cellulose capsules.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Scale HLV Clinical Formula Hair Vitamins — For the first week, participants will take 1 capsule in the morning and 2 capsules in the evening before food. From Week 2 onwards, participants will take 3 capsules daily in the evening before food.
  Arms: Intervention
Other: Placebo — For the first week, participants will take 1 capsule in the morning and 2 capsules in the evening before food. From Week 2 onwards, participants will take 3 capsules daily in the evening before food.
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy of Scale Media's HLV Clinical Formula Hair Vitamins on the health and appearance of hair, focusing on growth, volume, dullness, overall health, hair shedding, fullness, and strength. It is a randomized controlled trial with 50 female-at-birth participants experiencing self-perceived hair thinning.

ELIGIBILITY:
Inclusion Criteria:

* Female at birth, aged 35+.
* Self-perceived hair thinning and increased hair shedding for at least three months.
* Consistent hair care routine for at least one month prior.
* Willing to maintain hair care routine, diet, and refrain from new vitamins or supplements targeting hair growth during the study.
* Generally healthy without uncontrolled chronic diseases.

Exclusion Criteria:

* Hair loss conditions other than female pattern baldness.
* Pregnant, breastfeeding, or trying to conceive.
* Currently taking iron supplements or other hair growth treatments.
* Significant chronic conditions or planned medical procedures that interfere with protocol adherence.
* Recent chemical hair treatments or plans for such treatments during the study.
* Severe allergic reactions to the product's ingredients.
* Recent surgeries, major illnesses, or undergoing chemotherapy/radiotherapy.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-09-26 (Estimated); Study Completion 2024-09-26 (Estimated)

PRIMARY OUTCOMES:
Reduction in Hair Shedding | Baseline, Day 90, and Day 180
  Hair shedding will be measured through hair counts from the at-home comb test and hair health will be evaluated through expert dermatologist grading based on photos provided by participants.

SECONDARY OUTCOMES:
Improvement in Hair Health Perception | Baseline, Day 30, Day 60, Day 90, Day 120, Day 150, and Day 180
  Participants' perceptions of the product's effect on overall hair health, including volume, dullness, fullness, and strength, will be evaluated through self-reported questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The plan includes sharing individual participant data (IPD) collected during the study. The data to be shared includes de-identified individual participant data that underlie the results reported in the publication, including text, tables, figures, and appendices.